CLINICAL TRIAL: NCT04177706
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy of Ketamine for the Treatment of Concurrent Opioid Use Disorder and Major Depressive Disorder
Brief Title: Ketamine for the Treatment of Opioid Use Disorder and Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Jones, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00091292; K12DA031794 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Depression; Opioid-use Disorder; Opioid Abuse
Keywords: Ketamine
MeSH Terms: conditions — Depression; Opioid-Related Disorders | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Ketamine) (Experimental)
  Interventions: Drug: Ketamine Hydrochloride
- Group B (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Participants receiving the active study medication will receive 60 mg ketamine twice per week for four weeks under clinical supervision.
  Arms: Group A (Ketamine)
Drug: Placebo — Participants receiving the placebo study medication will receive saline twice per week for four weeks under clinical supervision.
  Arms: Group B (Placebo)

SUMMARY:
The purpose of the study is to examine whether an investigational medication called ketamine is able to improve treatment outcomes for concurrent opioid addiction and depression when used in conjunction with buprenorphine treatment. Study medications will be delivered twice per week for four weeks. If you are eligible and you decide to enroll in the study, your participation will last approximately 8 weeks, or 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 to 65 years old.
2. Able to provide informed consent.
3. Meet DSM-5 criteria for Major Depressive Disorder, without psychotic features.
4. Score at least 20 on the Montgomery-Asberg Depression Rating Scale.
5. Fulfill a minimum of 4 of 11 current opioid use disorder criteria by DSM-5.
6. Have used opioids illicitly at least once in the past month.
7. Subjects must be on standard of care pharmacotherapy for OUD (buprenorphine) for at least one month.
8. Subjects taking other psychotropic medications (e.g. anti-depressants or non benzodiazepine anxiolytics) must be maintained on a stable dose for at least four weeks before study initiation.
9. Subjects must be considered to have treatment-refractory MDD as evidenced by failure or only partial response to treatment with at least two standard of care pharmacotherapy antidepressants.
10. Must consent to random assignment to intranasal ketamine or placebo control.

Exclusion Criteria:

They are considered an immediate suicide risk (by Columbia Suicide Severity Rating Scale of 4 or greater, a history of a suicide attempt in the past year, or by clinician judgment) or felt to be likely to require hospitalization during the course of the study.

2. They have a self-reported history of illicit ketamine use, or baseline urine drug testing positive for ketamine.

3. They are in acute opioid withdrawal (as evidenced by a score of 5 or above on the Clinician Opioid Withdrawal Scale). These subjects will be referred for clinical detoxification and pharmacotherapy induction. Subjects may be re-assessed for study eligibility after one month of treatment with a standard of care OUD pharmacotherapy.

4. Subjects who meet DSM-5 criteria for current bipolar disorder. 5. Subjects who meet DSM-5 criteria for current or history of psychotic spectrum disorders.

6. Women who are pregnant or nursing. 7. Subjects with current hypertension as defined by a systolic blood pressure (SBP) >140 mmHg or a diastolic blood pressure (DBP) >90 mmHg.

8. Subjects with a self-reported history of delirium for any cause. 9. A history of allergic or other adverse reaction to ketamine. 10. Clinically significant abnormal laboratory values, physical exam findings or self-reported medical conditions for which a transient increase in blood pressure could be significantly detrimental (e.g. glaucoma, brain aneurysms, cardiovascular disease, or end-stage renal disease).

11. Electrocardiogram (ECG) findings (obtained within thirty days prior to randomization) of tachycardia, prior myocardial infarction, myocardial ischemia, or aberrant conduction).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Ketamine) | Group B (Placebo)
Started | 11 | 10
Completed | 6 | 5
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Ketamine) | Group B (Placebo) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Full Range); unit: years] | 35 [21 to 49] | 37 [29 to 58] | 36 [21 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Individuals Completing Informed Consent
Description: Primary outcomes will be 1) the percentage of individuals completing informed consent out of the number of individuals eligible on the initial screening.
Time Frame: Actual time frame of: 23 months.
Population: Outcomes will be cumulatively assessed from the time that the first participant is screened through the time that the last participant completes informed consent. There is only a single cohort (single arm/group) until randomization, which happens at the first interventional visit. Actual time frame of: 23 months.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Individuals Completing Informed Consent: Percentage of individuals completing informed consent out of the number of individuals eligible on the initial screening.
Arm/Group | Percentage of Individuals Completing Informed Consent
Number analyzed (Participants) | 153
Participants | 34

2. Primary Outcome: Percentage of Individuals Completing the Full Protocol
Description: The other primary outcome will be the percentage of individuals that complete informed consent which complete the full interventional protocol.
Time Frame: Actual time frame 23 months.
Population: There is only a single cohort (single arm/group) until randomization, which happens at the first interventional visit.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Individuals Completing the Full Study Treatment Protocol: Percentage of individuals completing the full study treatment protocol out of the total number that completed the informed consent.
Arm/Group | Percentage of Individuals Completing the Full Study Treatment Protocol
Number analyzed (Participants) | 34
Participants | 11

3. Secondary Outcome: Change in Depression Severity
Description: Secondary outcomes will include changes in depression severity (as measured on the Montgomery-Asberg Depression Rating Scale), which will be calculated as a change from baseline to 4 weeks (8th interventional visit). Montgomery Asberg Depression Rating Scale (MADRS; Montgomery, 1979). The MADRS is a clinician administered, 10-item questionnaire of depression severity. The total score ranges from 0-60, with scores of 0-6 considered normal (non-depressed), 7-19 indicative of mild depression, 20-34 indicative of moderate depression, and 35-60 indicative of severe depression. Individuals scoring 20 or higher on the MADRS will be included in the study. The MADRS evaluates the following symptoms of depression: 1) clinical appearance of sadness, 2) self-reported sadness, 3) inner tension, 4) reduced sleep, 5) reduced appetite, 6) concentration difficulties, 7) lassitude, 8) inability to feel, 9) pessimistic thought process, and 10) thoughts of suicide.
Time Frame: Baseline through 4-week interventional visits (8th interventional visit).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A (Ketamine) | Group B (Placebo)
Number analyzed (Participants) | 6 | 5
score on a scale | 30 (2.8) | 10.8 (14.1)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Group A (Ketamine) | Group B (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT04177706/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04177706/ICF_001.pdf